CLINICAL TRIAL: NCT06830616
Title: Acute Concussion Management in Emergency Medicine with 7T MRI: a Feasibility Study
Acronym: ACME-7T
Status: Not yet recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: INGN24HS153
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury (TBI); Concussion, Initial Encounter
Keywords: concussion; 7T MRI; head injury; mildTBI; MRI brain
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients who have completely recovered from concussion: Recovery from concussion will be assessed at 25 +/- 3 days using a validated symptom score, the Post Concussion Symptom Scale (PCSS). This group will have a PCSS = 0.
  Interventions: Diagnostic Test: 7T MRI brain
- Patients who have ongoing symptoms from concussion: Recovery from concussion will be assessed at 25 +/- 3 days using a validated symptom score, the Post Concussion Symptom Scale (PCSS). This group will have a PCSS > 10.
  Interventions: Diagnostic Test: 7T MRI brain

INTERVENTIONS:
Diagnostic Test: 7T MRI brain — A very detailed MRI scan of the brain using a 7T MRI scanner.

SUMMARY:
The goal of this observational study is to learn about the brain imaging changes associated with concussion using a very detailed (7T) MRI scanner.

To do this, the investigators will study 7T MRI brain imaging in patients aged 18-40 who present to the Emergency Department within 96 hours of a head injury. Patients will be eligible if they have had a normal CT brain as part of their usual care.

The investigators will compare brain imaging from patients who have completely recovered from an episode of concussion to patients who still have significant symptoms at approximately 28 days after a head injury.

The study attempts to answer the following questions:

1. Do patients with ongoing symptoms after concussion show greater 7T MRI brain imaging evidence of changes to the blood vessels at approximately 28 days after their injury in comparison to patients who have recovered fully?
2. Do patients with ongoing symptoms after concussion show greater 7T MRI brain imaging evidence of changes in brain signaling pathways at approximately 28 days after their injury, in comparison to patients who have recovered fully?

DETAILED DESCRIPTION:
Evaluation of symptoms will be conducted at presentation in the Emergency Department and at 25 +/- 3 days after head injury. This will be assessed using 2 validated questionnaires: the Neurological Assessment Questionnaire (NAQ) and the Post Concussion Symptom Scale (PCSS).

Lifetime incidence of concussion will be assessed at 7T MRI using the a modified version of the Brain Injury Screening Questionnaire (BISQ).

Information will also be collected regarding painkiller use, anticoagulation, return to work, and any related further unscheduled care admissions or CT head imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Isolated head trauma
2. Initial review within 96h of injury
3. No acute findings on CT head
4. Aged 18-40 years

Exclusion Criteria:

1. Patient unable to give informed consent
2. Patient unable to speak and understand English
3. Patients where alternative diagnosis cannot be excluded
4. Polytrauma
5. Contra-indication to MRI
6. BMI >40 or unable to comfortably lie on MRI scanner
7. Pregnant
8. Major confounding neurological disease e.g Multiple sclerosis, Stroke, Parkinson's Disease.
9. Patient participation in other research studies concurrently

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited from the Emergency Department at the Queen Elizabeth University Hospital, NHS Greater Glasgow and Clyde.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Microvascular Pathology (Blood Vessel Changes) on 7T MRI brain | 28 +/- 14 days from head injury
  To explore whether patients with ongoing symptoms after a concussion show greater 7T MRI brain imaging evidence of microvascular pathology (blood vessel changes) at 28 (± 14) days after their injury in comparison to patients who have recovered fully.

SECONDARY OUTCOMES:
Changes in Brain Signalling Pathways on 7T MRI | At 28 +/- 14 days from head injury
  To explore whether patients with ongoing symptoms after concussion show greater 7T MRI brain imaging evidence of ongoing metabolic disturbance in brain signalling pathways at 28 (± 14) days after their injury, in comparison to patients who have recovered fully.

IPD SHARING:
Plan to Share IPD: No